CLINICAL TRIAL: NCT05198336
Title: Immunogenicity of an Inactivated COVID-19 Vaccine for Prevention of COVID-19 in Population Aged 3-11 Years
Brief Title: Immunogenicity of an Inactivated COVID-19 Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-MA4007-SD
Record Dates: First submitted 2022-01-19; First posted 2022-01-20 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group of children aged 3-5 years old (Experimental): 200 subjects aged 3-5 years old who have received two doses of inactivated COVID-19 vaccine(CoronaVac) manufactured by Sinovac Research & Development Co., Ltd and is currently 28-42 days after the second dose
  Interventions: Biological: Inactivated COVID-19 Vaccine
- Experimental Group of children aged 6-11 years old (Experimental): 200 subjects aged 6-11 years old who have received two doses of inactivated COVID-19 vaccine(CoronaVac) manufactured by Sinovac Research & Development Co., Ltd and is currently 28-42 days after the second dose
  Interventions: Biological: Inactivated COVID-19 Vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 Vaccine — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac

SUMMARY:
This study is an open phase 4 clinical trial of an inactivated COVID-19 vaccine (CoronaVac) manufactured by Sinovac Research and Development Co., Ltd. The purpose of this study is to evaluate the immunogenicity of the CoronaVac in healthy children aged 3-11 years old.

DETAILED DESCRIPTION:
This study is an open phase 4 clinical trial to evaluate the immunogenicity of an inactivated COVID-19 vaccine(CoronaVac)in healthy children aged 3-11 years old.A total of 400 healthy subjects who have received two doses of inactivated COVID-19 vaccine(CoronaVac) manufactured by Sinovac Research & Development Co., Ltd and is currently 28-42 days after the second dose will be enrolled, including 200 subjects aged 3-5 years and 200 subjects aged 6-11 years old.All of subjects will be collected 3ml venous blood to evaluate the immunogenicity of the CoronaVac.

ELIGIBILITY:
Inclusion Criteria:

* Have received two doses of inactivated COVID-19 vaccine(CoronaVac) manufactured by Sinovac Research & Development Co., Ltd and is currently 28-42 days after the second dose;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (for subjects aged 8 years, both subjects and guardians need to sign the informed consent form);
* The subjects and their legal guardians voluntarily participate the study and comply with the study procedure to collect 3ml venous blood;
* Proven legal identity.

Exclusion Criteria:

* Haven't received two doses of inactivated COVID-19 vaccine(CoronaVac);
* Have received COVID-19 vaccines from other manufacturers;
* The interval between blood collection and the second dose is less than 28 days or more than 42 days;
* The subjets and their legal guardians can't cooperate to complete 3ml venous blood collection.
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 395 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-Seropositivity rate of the neutralizing antibody to SARS-CoV-2 | Day 28(+14 days) after the second dose of vaccine
  Seropositivity rate of the neutralizing antibody day 28(+14 days) after the second dose of vaccine
Immunogenicity index-GMT of the neutralizing antibody to SARS-CoV-2 | Day 28(+14 days) after the second dose of vaccine
  GMT of the neutralizing antibody to SARS-CoV-2 day 28(+14 days) after the second dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xu, Principal Investigator — Shandong Provincial Center for Disease Control and Prevention
Locations (1):
- Rushan City Center for Disease Control and Prevention, Weihai, Shandong, China